CLINICAL TRIAL: NCT02714751
Title: Evaluation of an Informative Intervention to the ICU Team About the Presence of Asynchronies in Mechanically Ventilated Patients: Effect Over Incidence Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Lluis Blanch, PhD, Corporacion Parc Tauli
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: CIR2015/057
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Asynchronies

ARMS (2):
- Observational group (No Intervention)
- Group after information intervention (Other): Control group after daily information to healthcare team
  Interventions: Behavioral: Daily asynchronies information

INTERVENTIONS:
Behavioral: Daily asynchronies information
  Arms: Group after information intervention

SUMMARY:
Mechanical ventilation (MV) if a life-support treatment for critically ill patients that can develop adverse effects. Patient-ventilator asynchronies can be present from the beginning of MV, it can be associated with poor outcome and it can develop clinical changes. The aim of this study is to evaluate if the knowledge of the presence of asynchronies by the healthcare team can help to reduce its incidence, improving outcomes of critically ill patients.

A prospective, single-center, before and after study will be conducted in the ICU of Hospital de Sabadell. The study will have 2 phases: a first observational period where the incidence of asynchronies will be assessed, and a second period where a daily information of the presence of asynchronies to the healthcare team will be done with the aim to reduce the incidence.

A continous record of asynchronies and clinical variables will be done during ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation < 24 hours.
* > 18 years-old

Exclusion Criteria:

* > 24 hours of invasive mechanical ventilation at admission.
* <48 hours of data collected
* Informed consent not obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2016-03; Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Incidence of asynchronies | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Tauli, Sabadell, Spain